CLINICAL TRIAL: NCT05567081
Title: Efficacy of Ultrasound-Guided Deep Perineural Platelet Rich Plasma Versus Corticosteroid Injection in Patients With Ulnar Neuropathy at Elbow, a Comparative Study
Brief Title: Efficacy of Ultrasound-Guided PRP Versus Corticosteroid Injection in Patients With Ulnar Neuropathy at Elbow
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hajar Anwer Elnagar, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34743/6/21
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Ulnar Neuropathy at Elbow
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): 3 cm of autologous platelet rich plasma injected once around the thickest part of ulnar nerve.
  Interventions: Drug: PRP
- Corticosteroid group (Experimental): Triamcinolone Acetonide 40mg/mL (1ml) mixed with 1ml lidocaine hydrochloride injected once around the thickest part of ulnar nerve.
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — Deep perineural injection with 1cm corticosteroid mixed with 1ml lidocaine hydrochloride.
  Other Names: Epirelefan 40 mg
  Arms: Corticosteroid group
Drug: PRP — Deep perineural injection with 3ml PRP at the thickest part of the ulnar nerve.
  Arms: PRP group

SUMMARY:
This study was be performed on 60 patients with ulnar neuropathy at elbow diagnosed clinically and by electrophysiology and/or ultrasonography selected from Physical medicine, Rheumatology & Rehabilitation Department, Faculty of Medicine, Tanta University.

Patients were be randomly divided into 2 groups:

Group I: will undergo a single ultrasound-guided deep perineural injection with 3ml PRP at the thickest part of the ulnar nerve. PRP will be prepared by PRP method.

Group II: will undergo a single ultrasound-guided deep perineural injection with 1ml corticosteroid (triamcinolone acetonide, 40mg/mL) mixed with 1ml lidocaine hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulnar neuropathy at elbow diagnosed clinically and by electrophysiology and/or ultrasonography.

Exclusion Criteria:

1. Patients with severe ulnar neuropathy at elbow according to Gu's classification. 15
2. Brachial plexopathy, peripheral neuropathy, and cervical radiculopathy.
3. History of recent elbow trauma or operation.
4. Malignant neoplasm.
5. Pregnancy.
6. Bleeding Disorders.
7. Factors affecting nerve healing process e.g., tobacco use and systemic corticosteroid administration.
8. Contraindications for PRP injection:

   1. Significant renal or hepatic dysfunction.
   2. Critical thrombocytopenia.
   3. Hemodynamic instability.
   4. Septicemia.
   5. Local infection at the site of the procedure.
   6. Consistent use of nonsteroidal anti-inflammatory drugs within the last two weeks.
   7. Local injection at the suspected treatment site within the last month.
   8. Recent fever or illness.
   9. Hemoglobin level <10 g/dL.
   10. Platelet dysfunction disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Change in ultrasound cross sectional area of ulnar nerve at elbow after injection | 1, and 3 months after injection
Change in nerve conduction parameters of ulnar nerve at elbow after injection | 1 and 3 months after injection
  Change in ulnar nerve conduction velocity and CMAP across elbow.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided